CLINICAL TRIAL: NCT02622464
Title: Innovative Treatment for Scarred Vocal Cords by Local Injection of Autologous Stromal Vascular Fraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-01
Record Dates: First submitted 2015-11-19; First posted 2015-12-04 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2018-09

CONDITIONS: Dysphonia
MeSH Terms: conditions — Dysphonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- micro injection of SVF in vocal cords (Experimental): micro injection of Stromal Vascular Fraction extracted from autologous adipose tissue in vocal cords
  Interventions: Other: micro injection of SVF in vocal cords

INTERVENTIONS:
Other: micro injection of SVF in vocal cords

SUMMARY:
Post-operative scarring on vocal cords is responsible for disorders of the vibration of the lining to the original dysphonia can be troublesome for the patient both in his private and professional life. There is no currently codified treatment for this type of situation and no therapeutic antifibrotic has been effective. Cell therapy is a promising new approach.After a liposuction and removing of mature adipocytes (40 to 60%), the remaining cells called stromal vascular fraction (SVF) could be isolated. SVF consists of a heterogeneous cell population including multipotent stem cells similar to mesenchymal stem cells present in bone marrow. The investigators hypothesis is that the trophic and antifibrotic properties of SVF could benefit patients with vocal cords scarring responsible for dysphonia.

ELIGIBILITY:
Inclusion Criteria:

* Vocal Difficulties felt as crippling (VHI > 60/120)
* Presence of scar hurts of the caused vocal cords is by the initial surgery (micro-laryngoscopy in suspension with or without laser) or by a congenital pathology of glottidis sulcus
* Scar Aspect of vocal cords judged on a stroboscopic examination
* Delay of at least 1 year with regard to the initial surgery

Exclusion Criteria:

* Patients refusing the speech therapy
* Patients operated for a malignant lesion or in malignant potential serious dysplasia of the scar vocal cord
* Contraindication in the anesthesia
* Patients under anti-coagulants
* Patients presenting disorders of the coagulation
* Active infectious diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

PRIMARY OUTCOMES:
feasibility of Stromal Vascular Fraction injection injected in vocal cords | 13 months
  feasibility will be assessed by observation of the immediate volumizing effect on the edge free of the vocal cord appreciated on the video document
safety will be assessed by the absence of related events related to stromal vascular fraction injection injected in vocal cords | 13 months
  safety of Stromal Vascular Fraction injection injected in vocal cords

SECONDARY OUTCOMES:
efficiency of SVF injection for the treatment of scarred vocal cords with improved instrumental objective characteristics of the voice of the operated patients | 13 months
  efficiency of SVF injection will be assessed by visual analysis of the vocal cord vibration appreciated by vidéolaryngostroboscopy
efficiency of SVF injection for the treatment of scarred vocal cords with improved instrumental objective characteristics of the voice of the operated patients | 13 months
  efficiency will be assessed by the questionnaire Voice Handicap Index 30 (Jacobson)

CONTACTS AND LOCATIONS:
Overall Officials: Antoine GIOVANNI, MD, Principal Investigator — assistance publique hôpitaux de marseille; catherine GEINDRE, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assisitance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Mattei A, Bertrand B, Jouve E, Blaise T, Philandrianos C, Grimaud F, Giraudo L, Aboudou H, Dumoulin C, Arnaud L, Revis J, Galant C, Velier M, Veran J, Dignat-George F, Dessi P, Sabatier F, Magalon J, Giovanni A. Feasibility of First Injection of Autologous Adipose Tissue-Derived Stromal Vascular Fraction in Human Scarred Vocal Folds: A Nonrandomized Controlled Trial. JAMA Otolaryngol Head Neck Surg. 2020 Apr 1;146(4):355-363. doi: 10.1001/jamaoto.2019.4328. PMID 32053141